CLINICAL TRIAL: NCT00543101
Title: A Randomized, Controlled Trial to Evaluate the Efficacy of Substituting Darunavir/Ritonavir (DRV/r) for Dual-boosted Protease Inhibitors in Individuals With Virologic Suppression for at Least 12 Weeks
Brief Title: Efficacy Study of Substitution of Darunavir/Ritonavir (DRV/r) for Dual-boosted Protease Inhibitors
Acronym: DVD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-142
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Results first posted 2010-08-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; darunavir; Protease inhibitors; Dual boosted; Treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch to DRV/r (Active Comparator): Switch to DRV/r at a dose of 600/100 BID for 48 weeks
  Interventions: Drug: Darunavir (DRV/r)
- Continue on Current Dual Boosted PI (Active Comparator): Continue on current dual boosted PI until week 24. At week 24, participants will be allowed to cross over to the DRV/r arm provided that they have maintained virologic suppression (< 400 copies/ml) for the first 24-weeks of the study and are followed for an additional 24 weeks
  Interventions: Drug: continue on current dual boosted PI

INTERVENTIONS:
Drug: Darunavir (DRV/r) — Switch to DRV/r at a dose of 600/100 BID for 48 weeks
  Arms: Switch to DRV/r
Drug: continue on current dual boosted PI — Continue on current dual boosted PI until week 24. At week 24, participants will be allowed to cross over to the DRV/r arm provided that they have maintained virologic suppression (< 400 copies/ml) for the first 24-weeks of the study and be followed for an additional 24 weeks
  Arms: Continue on Current Dual Boosted PI

SUMMARY:
This study will evaluate patients who have achieved virologic suppression (< 400 copies/mL) on any dual protease inhibitor (PI) combination, to determine whether patients can substitute both PIs with the single boosted PI darunavir given 600/100 ritonavir (RTV) twice daily (BID) and maintain comparable virologic suppression (% < 50 c/mL) for 24 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to determine if patients who have achieved virologic suppression (< 400 copies/mL) on any dual PI combination, can substitute both PIs with the single boosted PI darunavir given 600/100 rtv bid and maintain comparable virologic suppression (% < 50 c/mL) for 24 weeks. Randomized, non-blinded, multicenter, 48 week, controlled trial to assess the non-inferiority of substituting DRV/r for a dual boosted PI combination in patients with stable virologic suppression on a regimen containing a dual boosted PI combination plus at least one additional FDA-licensed antiretroviral agent from another class. Participants will be randomized (1:1) to one of the included treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Treatment with a stable antiretroviral regimen containing two protease inhibitors, one additional FDA-licensed agent from another class (except NNRTIs) and a boosting dosage of ritonavir (100 BID or QD) for at least 12 weeks prior to screening
* No plans to make any changes in HIV treatment regimen (other than those required by study) in the next 48 weeks.
* HIV-1 RNA < 400 copies/ml based on the most recent value done as part of routine care at least 12 weeks prior to screening; and < 400 at screening
* Any CD4 count is allowed
* Written informed consent to participate

Exclusion Criteria:

* Current regimen includes an NNRTI
* CDC Class C Illness diagnosed within 30 days of screening
* Lab abnormalities as defined by a standardized grading scheme based on the DAIDS table
* Any grade 3 or 4 toxicity with the following exceptions:

  * Pre-existing diabetes with glucose elevations ≥ grade 3
  * triglyceride or total cholesterol elevations ≥ grade 3
* Clinical or laboratory evidence of clinically significant liver impairment/dysfunction, disease or cirrhosis Note: Individuals co-infected with chronic hepatitis B or C will be allowed to enter the trial if their condition is clinically stable. Individuals diagnosed with acute viral hepatitis at screening will not be allowed to enroll during acute phase.
* Active substance abuse or significant psychiatric illness that in the opinion of the investigator might interfere with study compliance.
* Use of any investigational agents 30 days prior to screening
* Life expectancy < 6 months in the opinion of the investigator
* Prior use of darunavir or known allergy to any of the components of darunavir
* Breast feeding
* Female subject of childbearing potential not using effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last trial related activity.

Note: Hormonal based contraception may not be reliable when taking darunavir, therefore to be eligible for this study, women of childbearing potential who may have vaginal intercourse should either:

1. Use a double barrier method to prevent pregnancy (i.e., using a condom with either a diaphragm or cervical cap) Or
2. Use hormonal based contraceptives in combination with a barrier contraceptive (i.e., male condom, diaphragm, cervical cap or female condom) Or
3. Use an intra uterine device (IUD) in combination with a barrier contraceptive (i.e., male condom, diaphragm, cervical cap or female condom) Or
4. Be non-heterosexually active, practice sexual abstinence or have a vasectomized partner (confirmed sterile).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin J Cohen, MD, MSc, Principal Investigator — CRI
Locations (5):
- United States (5):
  - Spectrum Medical Group, Phoenix, Arizona
  - AIDS Healthcare Foundation, Los Angeles, California
  - Orlando Immunology Center, Orlando, Florida
  - Community Research Initiative of New England, Boston, Massachusetts
  - Albany Medical Center, Albany, New York

REFERENCES:
- See also: Web page of CRI, the nonprofit research group sponsoring the study — http://www.crine.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five multicenter sites were used these included medical and research clinics.
Groups:
- Continue on Current Dual Boosted PI: This is the control group. Subjects in this arm stay on their current regimen - a dual boosted PI combination.
Period: Overall Study
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 46 [31 to 59] | 51 [36 to 64] | 50 [31 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Successful Virologic Suppression
Description: Amount of HIV RNA copies per ml blood collected from subjects as measured by the Ultra-sensitive HIV-1 PCR (Roche Cobas). Successful virologic suppression is defined as < 50 copies/ml blood. The result is the percentage of participants with successful virologic suppression.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI
Number analyzed (Participants) | 12 | 12
Percentage of Participants | 100 | 100

2. Secondary Outcome: Economic Impact of a Substitution of Dual Boosted PIs With DRV/r
Description: To assess the economic impact of DRV/r substitution for dual boosted PIs, we compared the average wholesale acquisition costs for the drugs in US Dollars ($) per month. The wholesale acquisition cost in US dollars ($) for each ART regimen was determined and the difference between the cost for the experimental and control groups was calculated and reported as US dollar savings per month.
Time Frame: 48 weeks
Measure: Number; unit: US dollars savings per month
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI
Number analyzed (Participants) | 12 | 12
US dollars savings per month | 217 | 0

3. Secondary Outcome: Lipid Fraction Results, Mean of the Change From Baseline to Week 24.
Description: We collected fasting total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides from all participants in both arms of the study. We calculated the differences between the values at week 24 and baseline for the participants in both arms. We reported the mean of the change from baseline to week 24.
Time Frame: baseline and 24 weeks
Measure: Number; unit: mg/dL
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI
Number analyzed (Participants) | 12 | 12
mg/dL
  Change in Total Cholesterol | -6 (NA) | 2
  Change in LDL-Cholesterol | -4 | 2
  Change in HDL-Cholesterol | -1 | 1
  Change in Triglycerides | -13 | 0

4. Secondary Outcome: Treatment Satisfaction (+3, Much More Satisfied Now to -3, Much Less Satisfied Now)
Description: Participants in the experimental arm completed treatment satisfaction questionnaires at 24 weeks, and the control arm at 48 weeks (24 weeks after mid-study crossover to boosted darunavir). The questionnaires used numeric satisfaction scales (+3 much more satisfied now to -3 much less satisfied now). We reported the median and ranges for each question for each study arm.
Time Frame: 24 weeks
Measure: Median (Full Range); unit: Units on a Scale (+3 to -3)
Groups:
- Crossover Week 48: At week 24 the dual PI arm subjects remaining undetectable, crossed over to the DRV/r arm and were followed for an additional 24 weeks.
Arm/Group | Switch to DRV/r | Crossover Week 48
Number analyzed (Participants) | 12 | 7
Units on a Scale (+3 to -3)
  How satisfied are your with your current treatment | 3 [0 to 3] | 2.5 [2 to 3]
  How satisfied are you with any side-effects | 2 [0 to 3] | 2.5 [2 to 3]
  How convenient is your treatment | 3 [-1 to 3] | 3 [2 to 3]
  How well does your treatment fit your lifestyle | 3 [-1 to 3] | 3 [2 to 3]
  Would you recommend your treatment to someone else | 3 [0 to 3] | 2.5 [2 to 3]
  How likely are you to continue your treatment | 3 [0 to 3] | 2.5 [1 to 3]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over the course of the study (about 2 years)
Arm/Group | Switch to DRV/r | Continue on Current Dual Boosted PI
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/12
Other Adverse Events (participants affected / at risk) | 7/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to DRV/r (N=12) | Continue on Current Dual Boosted PI (N=12)
Abnormal Total Bilirubin (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bilirubin Grade 3 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Elevated Triglycerides (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to DRV/r (N=12) | Continue on Current Dual Boosted PI (N=12)
anal ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
bilateral ankle and pedal edema (Vascular disorders) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
coarse rhonchi bilaterally (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (General disorders) | 0 (0) | 1 (1)
decreased range of motion, left shoulder/arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dental (General disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
earache (Ear and labyrinth disorders) | 2 (2) | 0 (0)
elevated blood pressure, intermittent (Vascular disorders) | 1 (1) | 0 (0)
flu (Infections and infestations) | 0 (0) | 1 (1)
fractured sternum (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
intermittent tingling on tongue with metallic taste (Nervous system disorders) | 1 (1) | 0 (0)
intermittent numbness left face/tongue (Nervous system disorders) | 1 (1) | 0 (0)
left molar abscess (Infections and infestations) | 1 (1) | 0 (0)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
malaise (General disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nose fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
pubic region (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
recurrence of squamous cell carcinoma in situ-colorectal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
right arm pain (secondary to motor vehicle accident) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
right hip pain (secondary to motor vehicle accident) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
right knee pain (secondary to motor vehicle accident) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
symptoms of memory loss (Nervous system disorders) | 1 (1) | 0 (0)
worsening hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
worsening hypertension (Vascular disorders) | 1 (1) | 0 (0)
abscess posterior right thigh (Infections and infestations) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
abnormal liver function test (Hepatobiliary disorders) | 4 (6) | 4 (5)
anal fissure (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
asthmatic, bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
bilateral inguinal lymphadeopathy (Immune system disorders) | 0 (0) | 1 (1)
body aches (General disorders) | 1 (1) | 0 (0)
body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
broken wrist (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
contusion, right forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
creatinine (Renal and urinary disorders) | 1 (1) | 1 (2)
elevated cholesterol (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
elevated glucose (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
elevated triglycerides (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
eye irritation (Eye disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
headache (Vascular disorders) | 1 (1) | 1 (1)
herpes glands penis (Infections and infestations) | 0 (0) | 1 (1)
herpes simplex UPNI (HSV) on face (Infections and infestations) | 0 (0) | 1 (1)
herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
inflammation penis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 0 (0) | 1 (1)
lymphadenopathy (Immune system disorders) | 0 (0) | 1 (1)
meralgia paresthetica (Nervous system disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
neuropathic symptoms (Infections and infestations) | 1 (1) | 0 (0)
open wound, finger (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
periodontal disease (Infections and infestations) | 1 (1) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pulled hamstring (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
respiratory infection (Infections and infestations) | 2 (2) | 1 (2)
sebaceous cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
sore throat (Infections and infestations) | 1 (1) | 0 (0)
suprapubic abscess (Infections and infestations) | 1 (1) | 0 (0)
viral syndrome (Infections and infestations) | 0 (0) | 1 (2)
wrist sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The foremost problem was the small number of participants enrolled. By the time we were open for enrollment, most clinicians in the community had already switched their patients from dual boosted regimens to darunavir/ritonavir.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site Investigators (PIs) agree not to individually publish the results of the study. They may participate in a joint publication of the study results with the sponsor.